CLINICAL TRIAL: NCT02773511
Title: Multi-center Study on Surgical or Non-surgical Treatment for Children Type 1 Humeral Condyle Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Li Jin, Wuhan Union Hospital, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WuhanUH
Record Dates: First submitted 2016-05-13; First posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Treatment for Type I Humeral Condyle Fracture
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bone healing (Other): Bone healing in surgical or conservative treatment for children type 1 humeral condyle fracture
  Interventions: Procedure: Surgical treatment
- Fracture displacement (Other): Fracture displacement in surgical or conservative treatment for children type 1 humeral condyle fracture
  Interventions: Procedure: Surgical treatment

INTERVENTIONS:
Procedure: Surgical treatment — Closed reduction and Kirschner wire fixation

SUMMARY:
The study evaluates the effectiveness of surgical or non-surgical treatment for children type 1 humeral condyle fracture.Half of the participants receive surgical treatment and the other half receive non-surgical treatment

ELIGIBILITY:
Inclusion Criteria:

Children Type 1 humeral Condyle Fracture，Fracture displacement less than 2mm

Exclusion Criteria:

Other type humeral Condyle Fracture

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Fracture displacement rate | 1 months
Fracture healing rate | 3 years